CLINICAL TRIAL: NCT04803435
Title: Telemedicine Evaluation of Immunocompetent Adult Patients With Symptoms Suggestive of Acute Gastrointestinal Infection Compared With Face-to-face Medical Consultation in an Emergency Department: a Randomized Study of Diagnostic Accuracy
Brief Title: Telemedicine and Face-to-face Consultations Diagnostic Accuracy Comparison in Gastrointestinal Infection Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital Israelita Albert Einstein (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 36793220300000071
Record Dates: First submitted 2021-03-11; First posted 2021-03-17 (Actual); Last update posted 2022-02-11 (Actual); Status verified 2021-03

CONDITIONS: Gastrointestinal Infection
Keywords: Diarrhea; Telemedicine; Emergency Medical Services
MeSH Terms: conditions — Diarrhea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adult patients with acute gastrointestinal infection - telemedicine before face-to-face evaluation (Active Comparator): Adult patients who sought in person the screening of the Morumbi Emergency Care Unit of HIAE with symptoms suggestive of GECA (diarrhea with or without other symptoms of the digestive tract and infectious) who have undergone telemedicine consultation before face-to-face evaluation
  Interventions: Other: Telemedicine Consultation; Other: Face-to-face Consultation
- Adult patients with acute gastrointestinal infection - only face-to-face evaluation (Active Comparator): Adult patients who sought in person the screening of the Morumbi Emergency Care Unit of HIAE with symptoms suggestive of GECA (diarrhea with or without other symptoms of the digestive tract and infectious) who have only face-to-face evaluation
  Interventions: Other: Face-to-face Consultation

INTERVENTIONS:
Other: Telemedicine Consultation — Brief telemedicine consultation, blindedto subsequent face-to-face evaluation.
  Arms: Adult patients with acute gastrointestinal infection - telemedicine before face-to-face evaluation
Other: Face-to-face Consultation — Direct face-to-face evaluation (without telemedicine consultation before).

SUMMARY:
Acute gastroenterocolitis (GECA) in healthy adults is a frequent cause of looking for medical care in emergency care units and most cases are aimed at etiology viral infection or food toxin, being generally self-limited with good prognosis and only need for treatment with behavioral measures and use of medications for relief symptomatic. Anamnesis is the main resource for the diagnosis and stratification of GECA severity and is infrequent alterations of physical examination and complementary examinations without association with symptoms of alert. Telemedicine has become a resource that allows easier and faster access to medical evaluation, with low cost and rational use of resources. Virtual emergency care is part of Hospital Israelita Albert Einstein (HIAE) institutional routine and there is a large number of consultations whose final diagnosis was GECA. It is not known whether the accuracy of diagnosis of GECA by telemedicine is not inferior to the diagnosis by face-to-face evaluation, considered the Golden pattern. The aim of the study is compare the diagnostic accuracy of GECA by telemedicine with that of face-to-face care. It is a prospective randomized study with a population of adult patients who sought in person the screening of the Morumbi Emergency Care Unit of HIAE with symptoms suggestive of GECA (diarrhea with or without other symptoms of the digestive tract and infectious). Patients whose screening will be excluded of nursing directed for immediate evaluation in the emergency room and patients with dysfunctions organisms or immunosuppression. Patients who accept and sign the informed consent form will be randomized into 2 groups: A) immediate face-to-face evaluation; B) evaluation initially by telemedicine and sequentially at face-to-face evaluation. In both cases, the ICD diagnostics will be compiled and grouped according to clinical significance and will be the primary outcome of the study. Service time, exams requested, guidelines, prescription and destination will also be analyzed. Patients and doctors who undergoing group B assessment will be blinded to the telemedicine assessment data.

DETAILED DESCRIPTION:
The face-to-face assessment will be carried out by the local UPA medical and assistance team and the assessment by telemedicine by the fixed medical team of the HIAE service responsible for urgency / emergency. Both in face-to-face evaluation, as well as telemedicine, clinical data, final diagnosis, destination, total time of care, guidance and prescription will be computed. In the face-to-face evaluation, complementary exams and medications received in situ were computed. Final diagnoses will receive nomenclature according to the International Statistical Classification of Diseases and Problems Health-Related - ICD 10 (institutional medical record requirement - Cerner) and will be grouped according to equivalence of syndromic diagnosis. The diagnosis of the face-to-face assessment is made according to protocols based on extensive medical literature and approved by the institutional clinical staff, being representative of current medical practice and will be considered the gold standard diagnosis. Patients evaluated by telemedicine will be blinded to the diagnosis, recommended destination, guidelines and prescription performed by the medical team. UPA doctors will be blind to the doctor's assessment telemedicine and telemedicine doctors will not have access to the data obtained in the screening.

ELIGIBILITY:
Inclusion Criteria:

* Age> 18 years
* Symptoms present less than 7 days.
* Without the use of antibiotics in last 30 days prior to the onset of symptoms.
* No trips abroad in the last 15 days prior to the onset of symptoms.
* Presence of more than three episodes of watery diarrhea in the last 24 hours with or without symptoms related to the infection (fever 38oC, chills, sweating, myalgia, vomiting) that motivated / were looking for the Emergency Care Unit
* Signature of informed consent form

Exclusion Criteria:

* Return to the Emergency Care Unit due to maintenance or aggravation of the complaint
* Age> 65 years
* Diagnosis of chronic gastrointestinal diseases, gastritis with or without gastroesophageal reflux disease, previous diverticulitis, previous abdominal surgery, chronic colitis, inflammatory bowel diseases, food intolerances (gluten, lactose)
* Previous diagnosis of congestive heart failure, HIV / AIDS, active cancer, type I diabetes mellitus, use of any immunosuppressant
* Diarrhea chronic
* Patient with emergency room criteria by the nursing evaluation of the triage.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-02-20 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Accuracy of telemedicine diagnosis of adult patients with symptoms compatible with acute gastrointestinal infection | through study completion, an average of 1 year
  The patient will be evaluated by telemedicine and / or face-to-face consultation and at the end will receive the diagnosis, which will be assigned the ICD code. At the end, these ICDs will be grouped by the same clinical significance and will be compared between the two consultation methods (telemedicine versus face-to-face consultation).

SECONDARY OUTCOMES:
Time of medical care | through study completion, an average of 1 year
  Comparison of time (minutes) of medical care between telemedicine and face-to-face consultation.
Rate of indication for complementary exams | through study completion, an average of 1 year
  Comparison of rate (porcentage) of indication for complementary exams between telemedicine and face-to-face consultation.
Types of requested exams | through study completion, an average of 1 year
  Comparison of types of requested exams (porcentage) between telemedicine and face-to-face consultation.
Guidelines follow-up | through study completion, an average of 1 year
  Comparison of guidelines follow-up (porcentage) between telemedicine and face-to-face consultation.
Medical prescription | through study completion, an average of 1 year
  Comparison of medical prescription after completion of the service between telemedicine and face-to-face consultation.
Proposed destination after completion of the service | through study completion, an average of 1 year
  Comparison of proposed destination (percentage of discharge or hospitalization) after completion of the service between telemedicine and face-to-face consultation.

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo HS Cordioli, MD, Study Director — Telemedicine Department, Hospital Israelita Albert Einstein, Sao Paulo, Brazil